CLINICAL TRIAL: NCT04336644
Title: Continuous Versus Intermittent cARdiac Electrical moNitorinG
Acronym: CARING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202001147
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Torsades de Pointe Caused by Drug; Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Continuous patch monitoring system (Experimental): -Participants will receive standard of care treatment with either arsenic trioxide, ribociclib, or capecitabine. They will have continuous patch monitor system (BodyGuardian Mini Plus) applied on or prior to the first day of therapy and will receive at least 5 ECGs for comparison during the first 30 days of treatment.
  Interventions: Device: BodyGuardian Mini Plus

INTERVENTIONS:
Device: BodyGuardian Mini Plus — The BodyGuardian Mini Plus attaches to the upper chest of the patient through the use of an adhesive patch. ECG tracings are recorded continuously and sent to the linked smartphone and subsequently to a cloud server.
  Other Names: Continuous patch monitoring system

SUMMARY:
The purpose of this study is to validate the continuous patch monitoring system to evaluate cardiac arrhythmias in patients receiving drugs that can cause cardiac complications and compare the continuous patch system with standard electrocardiograms (ECGs).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL) and being initiated on standard of care arsenic trioxide OR Diagnosis of solid tumor and being initiated on standard of care capecitabine (alone or as part of combination treatment) OR Diagnosis of solid tumor and being initiated on standard of care ribociclib (alone or as part of combination treatment)
* At least 18 years of age.
* No allergy to adhesive patches.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Younger than 18 years of age
* Allergy to adhesive patches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of blinded, manual measurements of the ECGs to the patch monitor tracings as measured by the Bland-Altman Plot | Through Day 30
  * The Bland Altman plot provides a graphical method to compare the question of interest, namely that the measurements derived from the patch monitor are accurate in relation to the gold standard of the ECG.
  * Each QT measured from the tracing will be plotted against the difference in QT between the tracing and the 12-lead ECG. The acceptable difference between measurement techniques will be set at 5 ms (primary, strict threshold based on FDA recommendations) with a clinically acceptable difference of 15 ms (based on known variability in 12-lead ECG recordings).
Frequency of major arrhythmia occurrence | Through Day 30
  * The QT interval will be assessed every 4 hours for the first 5 days and then every 8 hours thereafter
Trajectories of QT prolongation | Through day 30
  * Will assess the QT interval every four hours for five days after drug initiation and after five days, the QTc will be assessed every 8 hours
  * With this data, the investigators will plot the QTc interval (Fridericia correction) over time and determine the time of expected peak effect. Outliers will be reviewed and verified manually.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Mitchell, M.D., FACC, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. We may also share your research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If your individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at your information.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Please email any proposals to jdmitchell@wustl.edu.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu